CLINICAL TRIAL: NCT01459523
Title: Optimizing Catheter Insertion Technique for Ultrasound-guided Continuous Peripheral Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Edward R. Mariano, Staff Physician, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21961
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Pain, Postoperative
Keywords: Peripheral Nerve Block; Perineural Catheter; Orthopedic Surgery; Ultrasound
MeSH Terms: conditions — Pain, Postoperative | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imaging technique (Active Comparator): In one substudy, subjects will be randomly assigned to either short axis or long axis target ultrasound imaging for perineural catheter insertion. The onset time of sensory anesthesia will be measured following local anesthetic bolus via the catheter.
  Interventions: Procedure: Short axis ultrasound; Procedure: Long axis
- Catheter location (Active Comparator): In another substudy, subjects will be randomly assigned to receive their perineural catheters either proximally or distally along the same target nerve or plexus.
  Interventions: Procedure: Proximal placement; Procedure: Distal placement

INTERVENTIONS:
Procedure: Proximal placement — Subjects assigned to this group will have their perineural catheter placed in a proximal position (higher up in the arm or leg) with ultrasound guidance. The onset time of sensory anesthesia will be measured following local anesthetic bolus via the catheter.
  Other Names: Perineural catheter; Ultrasound; Catheter placement technique
  Arms: Catheter location
Procedure: Short axis ultrasound — Subjects assigned to this group will have the target nerve or plexus identified in short axis (cross-section) using ultrasound. Perineural catheter insertion will be performed in-plane. The onset time of sensory anesthesia will be measured following local anesthetic bolus via the catheter.
  Other Names: Perineural catheter; Ultrasound; Catheter placement technique
  Arms: Imaging technique
Procedure: Long axis — Subjects assigned to this group will have the target nerve or plexus identified in long axis (longitudinal) using ultrasound. Perineural catheter insertion will be performed in-plane. The onset time of sensory anesthesia will be measured following local anesthetic bolus via the catheter.
  Other Names: Perineural catheter; Ultrasound; Catheter placement technique
  Arms: Imaging technique
Procedure: Distal placement — Subjects assigned to this group will have their perineural catheter placed in a distal position (further down in the arm or leg) with ultrasound guidance. The onset time of sensory anesthesia will be measured following local anesthetic bolus via the catheter.
  Other Names: Perineural catheter; Ultrasound; Catheter placement technique
  Arms: Catheter location

SUMMARY:
Continuous peripheral nerve blocks (CPNB; also known as "perineural" catheters) provide target-specific pain control for a variety of surgeries. There has been increasing interest in the use of ultrasound guidance for regional anesthesia, and many techniques using ultrasound alone for perineural catheter insertion have been described. Catheters may be placed at various points along the brachial plexus (for upper extremity procedures) or in proximity to the femoral and/or sciatic nerve (for lower extremity procedures). To date, the optimal ultrasound scanning technique, catheter insertion endpoint, catheter placement location per indication, for the majority of ultrasound-guided continuous peripheral nerve blocks remain unknown. This study will help provide important information related to optimal ultrasound scanning techniques and will help identify ways to improve the success rates, onset times, and analgesic effectiveness of these techniques for real patients undergoing surgical procedures.

DETAILED DESCRIPTION:
Primary Aim: To determine if there is an optimal scanning technique for ultrasound-guided perineural catheter insertion that will result in the most accurate tip placement in proximity to the target nerve or plexus.

Secondary Aim: To determine if there is an optimal location for ultrasound-guided perineural catheter insertion along a target nerve or plexus that will result in maximum local anesthetic infusion benefits.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age;
* Undergoing unilateral, upper (at or distal to the elbow) or lower (hip or distal) extremity orthopedic surgery, with moderate-to-severe postoperative pain expected; and
* Desiring a continuous perineural catheter for postoperative analgesia.

Exclusion criteria:

* Patients who will have difficulty understanding the study protocol or caring for the infusion pump/catheter system; or
* Patients with any known contraindication to study medications, insulin-dependent diabetes mellitus, neuropathy of any etiology in the affected extremity;
* Patients with a contraindication to regional blockade (eg, clotting deficiency);
* Patients with any known acute or chronic hepatic or renal insufficiency or failure;
* Patients with any additional surgical site outside of the catheter-affected area (eg, iliac crest bone graft in addition to hand surgery);
* Patients with chronic opioid use (defined as daily use for more than 4 weeks prior to surgery) or active illicit substance abuse;
* Patient weighing < 40 kg;
* Pregnancy;
* Incarceration; or
* Inability to communicate with the investigators and hospital staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Onset time of sensory anesthesia | 30 minutes
  The primary outcome will be the onset time of sensory anesthesia in the target nerve distribution following injection of a local anesthetic bolus via the perineural catheter.

SECONDARY OUTCOMES:
Time for placement | 30 minutes
  A secondary outcome measure will be the time required to insert the perineural catheter using the technique or location assigned.
Postoperative pain | 1 day
  A secondary outcome will be the surgical pain experienced by subjects as assessed by a 0-10 scale (0=no pain; 10=worst pain imaginable) and amount of opioid medications consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Edward R Mariano, MD, MAS, Principal Investigator — VA Palo Alto Health Care System (VAPAHCS)
Locations (1):
- VA Palo Alto Health System, Palo Alto, California, United States

REFERENCES:
- [Background] Grant SA, Nielsen KC, Greengrass RA, Steele SM, Klein SM. Continuous peripheral nerve block for ambulatory surgery. Reg Anesth Pain Med. 2001 May-Jun;26(3):209-14. doi: 10.1053/rapm.2001.22256. PMID 11359219
- [Background] Mariano ER, Cheng GS, Choy LP, Loland VJ, Bellars RH, Sandhu NS, Bishop ML, Lee DK, Maldonado RC, Ilfeld BM. Electrical stimulation versus ultrasound guidance for popliteal-sciatic perineural catheter insertion: a randomized controlled trial. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):480-5. doi: 10.1097/AAP.0b013e3181ada57a. PMID 19920423
- [Background] Mariano ER, Loland VJ, Bellars RH, Sandhu NS, Bishop ML, Abrams RA, Meunier MJ, Maldonado RC, Ferguson EJ, Ilfeld BM. Ultrasound guidance versus electrical stimulation for infraclavicular brachial plexus perineural catheter insertion. J Ultrasound Med. 2009 Sep;28(9):1211-8. doi: 10.7863/jum.2009.28.9.1211. PMID 19710219
- [Background] Mariano ER, Loland VJ, Sandhu NS, Bishop ML, Lee DK, Schwartz AK, Girard PJ, Ferguson EJ, Ilfeld BM. Comparative efficacy of ultrasound-guided and stimulating popliteal-sciatic perineural catheters for postoperative analgesia. Can J Anaesth. 2010 Oct;57(10):919-26. doi: 10.1007/s12630-010-9364-7. Epub 2010 Aug 11. PMID 20700680